CLINICAL TRIAL: NCT02497326
Title: Comparative Study of Conventional and Topical Heparin Treatments in Second Degree Burn Patients for Burn Analgesia and Duration of Wound Healing
Brief Title: Heparin for the Treatment of Burn Wound Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Mustehsan Bashir, Associate professor of Plastic Surgery, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 84/RC/KEMU
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Second Degree Burns
Keywords: second degree burns; heparin; topical
MeSH Terms: interventions — bacitracin, polymyxin B drug combination; Heparin; Tramadol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Polyfax & Lignocain gel or silvazine cream (Active Comparator): Polyfax skin ointment plus Lignocain gel will be applied on superficial PTB area and silver sulphadiazine cream on deep PTB in morning and evening after wound wash
  Interventions: Drug: Polyfax & Lignocain gel or silvazine cream; Drug: Tramadol
- Topical heparin (Experimental): Heparin solution (5000 IU/ml) will be sprinkled aseptically on burn surface twice a day for the first 2 days, by "#27" needle connected via drip set to the drip containing heparin aqueous saline. The dose will be reduced to 75% of day 1 on day 3 and 4 and to 50% on day 5. Administration of heparin saline solution will be in 3 cycles with 5-10 minutes interval.
  Interventions: Drug: Topical Heparin; Drug: Tramadol

INTERVENTIONS:
Drug: Polyfax & Lignocain gel or silvazine cream — olyfax skin ointment plus Lignocain gel will be applied on superficial PTB area and silver sulphadiazine cream on deep PTB in morning and evening after wound wash.
  Arms: Polyfax & Lignocain gel or silvazine cream
Drug: Topical Heparin — Heparin solution (5000 IU/ml) will be sprinkled aseptically on burn surface twice a day for the first 2 days, by "#27" needle connected via drip set to the drip containing heparin aqueous saline. The dose will be reduced to 75% of day 1 on day 3 and 4 and to 50% on day 5. Administration of heparin saline solution will be in 3 cycles with 5-10 minutes interval
  Arms: Topical heparin
Drug: Tramadol — IV Analgesic ( Inj. Tramadol 10mg/dose) will only be given to the patients (in both groups) having pain score >4, assessed 3 times a day by Numeric Visual Analogue scale (NVAS).

SUMMARY:
Pain Associated with partial thickness burns (PTB) is very severe and distressing for the patients.Topical conventional treatment of superficial PTB wounds includes application of polyfax skin ointment plus lignocain gel twice a day after wound wash while deep PTB are treated with silvazine cream twice a day and prepared for grafting if not healed within 3 weeks. Existing conventional therapy is un-comfortable and expensive for the patients. Search continues for a reliable, safe, cheap and effective treatment of burn.Topical use of heparin has been found effective in reducing pain associated with burn wounds. More over use of heparin topically in burn patients is easy to perform and cheap but at the moment, evidence of its effectiveness is weak. Current study is being conducted to verify clinical effectiveness of use of heparin in 2nd degree burns by comparing it with topical conventional treatment.

DETAILED DESCRIPTION:
Second degree or partial thickness burn (PTB) is most tricky variety to identify and treat, out of all four categories of burn (based on depth). It is further divided into superficial and deep partial thickness based on the depth of dermal injury. (1) Clinical criteria fulfilling all the points for each category i.e. Superficial PTB (SPTB) being reddish pink, bleed briskly (in <3sec) on pin prick, blanch with brisk return (in <2 sec) on pressure, blister formation and Deep PTB (DPTB) being mottled pink, delayed bleeding (in >3 sec) on pin prick, slow return (in >2 sec) on pressure, no blister, is most commonly used to differentiate both the sub-classes. Pain is hallmark of 2nd degree burns and is treated by topical and IV analgesics. Topical conventional treatment of superficial PTB wounds includes application of polyfax skin ointment plus lignocain gel twice a day after wound wash while deep PTB are treated with silvazine cream twice a day and prepared for grafting by normal saline dressings, if not healed within 3 weeks.

Current treatment for 2nd degree burn is complex, uncomfortable for the patient and expensive for the health systems (2,3) . Search continues for a reliable, safe, cheap and effective treatment of burn. Heparin has been used topically in burn patient and a protocol of topical heparin use has been introduced . It is believed that heparin helps in reducing pain associated with burns and duration of wound healing. (4) It is noted that the mechanism involved in heparin's action on the burn probably derives from its anti-inflammatory and angiogenic properties, stimulating tissue repair and re-epithelializing effects.(2) These actions do not depend on its well-known anticoagulant action. Burn analgesia by heparin is caused by inhibition of pro-inflammatory products which act on free nerve endings and cause pain. In this regard, isolated case reports continue to emerge, suggesting that heparin is able to promote tissue repair and inhibit inflammation in burn patients.(5) It has been shown in a study that out of total 58 patients, those in topical Heparin group demanded less analgesic medications in mg/day (11.83 ± 9.38) than Control group (33.35± 20.63) . It has been reported in another study that heparin applied topically for 5 days in 50 pediatric patients reduced healing time. (6) Indeed there are a number of reports of heparin being used, topically or systemically but there is a lack of effectively controlled studies in this area for clear conclusions to be drawn as to the efficacy of this approach.(7) As it is noted that already existing conventional therapy is un-comfortable and expensive for the patients, use of heparin topically in burn patients is easy to perform and cheap but at the moment, evidence of its effectiveness is weak. So rationale of the study is to verify clinical effectiveness of use of heparin in 2nd degree burns.

Objective:- To compare conventional treatment and topical heparin treatment in 2nd degree burn patients in terms of total consumption of analgesic medication and duration of wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender with age limits 14-60 years.
2. 2nd degree burn with Total burn surface area (TBSA) <20% (assessed by Wallace rule of nine) including front of chest and abdomen, upper limbs excluding hands and lower limbs excluding foot.
3. Flame and scald burn (on history).

Exclusion Criteria:

1. Third degree (painless, lathery eschar with no blanching) and Fourth degree burns (full thickness burn with exposed muscle, tendons or bones) as assessed clinically.
2. Chemical or electrical burn (on history).
3. Personal or family history of hemorrhagic diathesis, heparin intolerance, any medical illness causing bleeding episodes(e.g, Esophageal varices) or active bleeding from any site.
4. History of Liver disease (Total Bilirubin <20umol/L, Alanine amino transferase <36u/L, Aspartate amino transferase <42u/L), or renal disorder (Serum Urea=20-40mg/dl, Serum Creatinine <1.2).

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Total consumption of Analgesic Medication | 5 days
  Total consumption of Analgesic Medication will be calculated as total of the amount of IV analgesics required (mg/day) by patient, for the first 5 days of treatment, taking day of admission as "day 0". IV Analgesic ( Inj. Tramadol 10mg/dose) will only be given to the patients having pain score >4, assessed 3 times a day by Numeric Visual Analogue scale (NVAS).
Duration of wound healing | From date of staring treatment until the date when ≥70% re-epithelialization of SPTB has occured upto 21 days
  Duration of Wound Healing in SPTB will be assessed by
  1) Noting down the days required for the wound to re-epithelialize ≥70% . The number of day when ≥70% re-epithelialization has occured in SPTB will be noted taking day of starting treatment as 'day zero'
Duration of wound healing | Date on Twenty first day after starting treatment untill the date when DPTB ready for skin grafting
  Duration of Wound Healing in DPTB will be assessed by noting down days required for the wound to be ready for grafting in taking day 21 after staring treatment as "day 0" Wound will said to be ready for skin grafting if completely (100%) covered by granulation tissue with epithelialized margins.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Bashir, Principal Investigator — King Edward Medical University
Locations (1):
- Department of Plastic Surgery, Mayo Hospital, King Edward Medical University, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Klein MB. Thermal,chemical and electrical injuries In:Thorne CH et al.(ed.)Grabb and Smith's plastic surgery.7th ed. Philadelphia,Lippincott Williams & Wilkins;2014. p128 - 129. ISBN 978-1-4511-0955-9.
- [Background] Barretto MG, Costa Mda G, Serra MC, Afiune JB, Praxedes HE, Pagani E. [Comparative study of conventional and topical heparin treatments for burns analgesia]. Rev Assoc Med Bras (1992). 2010 Jan-Feb;56(1):51-5. doi: 10.1590/s0104-42302010000100016. Portuguese. PMID 20339787
- [Background] Klein MB, Hollingworth W, Rivara FP, Kramer CB, Askay SW, Heimbach DM, Gibran NS. Hospital costs associated with pediatric burn injury. J Burn Care Res. 2008 Jul-Aug;29(4):632-7. doi: 10.1097/BCR.0b013e31817db951. PMID 18535469
- [Background] Saliba MJ Jr. Heparin in the treatment of burns 2011". http://www.salibaburnsinstitute.org/ PROTOCOL.html.
- [Background] Ferreira Chacon JM, Mello de Andrea ML, Blanes L, Ferreira LM. Effects of topical application of 10,000 IU heparin on patients with perineal dermatitis and second-degree burns treated in a public pediatric hospital. J Tissue Viability. 2010 Nov;19(4):150-8. doi: 10.1016/j.jtv.2010.03.003. Epub 2010 Apr 20. PMID 20409713
- [Background] Venkatachalapathy TS. A comparative study of paediatric thermal burns treated with topical heparin and without heparin. Indian J Surg. 2014 Aug;76(4):282-7. doi: 10.1007/s12262-012-0674-6. Epub 2012 Oct 5. PMID 25278651
- [Background] Oremus M, Hanson MD, Whitlock R, Young E, Archer C, Dal Cin A, Gupta A, Raina P. A systematic review of heparin to treat burn injury. J Burn Care Res. 2007 Nov-Dec;28(6):794-804. doi: 10.1097/BCR.0b013e3181599b9b. PMID 17925636